CLINICAL TRIAL: NCT04802811
Title: A Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics, Pharmacodynamics of Oral SHR2150 in Healthy Subjects With Single Dose of SHR2150 in Healthy Subjects
Brief Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics ，Pharmacodynamics of Oral SHR2150 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SHR2150-I-103
Record Dates: First submitted 2021-03-10; First posted 2021-03-17 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-03

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment group A (Experimental)
  Interventions: Drug: SHR2150；Placebo
- Treatment group B (Experimental)
  Interventions: Drug: SHR2150；Placebo
- Treatment group C (Experimental)
  Interventions: Drug: SHR2150；Placebo
- Treatment group D (Experimental)
  Interventions: Drug: SHR2150；Placebo
- Treatment group E (Experimental)
  Interventions: Drug: SHR2150；Placebo

INTERVENTIONS:
Drug: SHR2150；Placebo — Single dose；SHR2150-dose 1 or Placebo-dose 1
  Arms: Treatment group A
Drug: SHR2150；Placebo — Single dose；SHR2150-dose 2 or Placebo-dose 2
  Arms: Treatment group B
Drug: SHR2150；Placebo — Single dose；SHR2150-dose 3 or Placebo-dose 3
  Arms: Treatment group C
Drug: SHR2150；Placebo — Single dose；SHR2150-dose 4 or Placebo-dose 4
  Arms: Treatment group D
Drug: SHR2150；Placebo — Single dose；SHR2150-dose 5 or Placebo-dose 5
  Arms: Treatment group E

SUMMARY:
The study is a randomized, Double-Blind, Placebo-Controlled study to evaluate the safety, tolerability and pharmacokinetics, pharmacodynamics of SHR2150.

will consist of 50 healthy subjects, 5 groups. The purpose of this part is to explore the safety, tolerability ,pharmacokinetics and pharmacodynamics of single doses of SHR2150 capsule in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Aged 18~45.
3. Body weight ≥ 50 kg for male; ≥ 45 kg for female, body mass index (BMI) between 18 to 28 kg/m2 ( Including boundary value) .
4. Vital signs, physical examination, laboratory results are within normal range or considered not clinically significant.
5. Female subjects (including partner) of childbearing potential must be using a medically acceptable form of birth control.

Exclusion Criteria:

1. Currently suffering from cardiovascular, liver, kidney, digestive, nervous, blood, thyroid or mental diseases.
2. Have severe infection, severe trauma or major surgical operations within 3 months. Plan to receive surgery during the trial and within two weeks after the end of the trial..
3. 12-ECG test have clinical significant abnormality or the QT interval (QTc) > 450 ms(male)/QTc)> 460 ms(male) or<300ms(female).
4. Screening for infectious diseases is positive (Including HBsAg, Anti-HCV, TPPA, Anti-HIV)
5. Suspected allergy to any ingredient in the study drug.
6. Have any drug that inhibits or induces liver metabolism within 1 month.
7. Any condition or disease that affects the absorption, metabolism, and/or excretion of the study drug judged by the investigator;
8. Treatment with immunosuppressant or interferon-containing drugs within 6 months of study drug administration;
9. Participated in clinical trials of any drug or medical device within 3 months before screening, or within 5 half-lives before screening;
10. Treatment with live(attenuated) vaccine within 2 months before taking the study drug or during the study or within 1 months after administration;
11. Had donated blood or blood transfusion≥ 200 mL within 1 months before taking the study drug or had donated blood or blood transfusion≥ 400 mL within 3 months prior to screening;
12. The average daily smoking ≥ 5 cigarettes within three months; the average daily alcohol intake in a month exceeds 15 g (15 g alcohol is equivalent to 450 mL beer or 150 mL wine or 50 mL low-alcohol);
13. Keep smoking, drinking alcohol or consuming caffeinated foods or beverages (more than 8 cups, 1 cup = 250 mL) 2 days before taking the study drug and during the study; and those who have special dietary requirements and cannot follow the unified diet;
14. History of drug abuse , drug dependence or drug screening test is positive;
15. Pregnant or lactating women;
16. Other conditions that the investigator believes the subject is not suitable.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of treatment-related adverse events as assessed by CTCAE v5.0. | 9 DAYS for Group A.B.C.D.E

SECONDARY OUTCOMES:
Pharmacokinetic parameters of SHR2150, , main metabolite and identified major metabolites in plasma ：[AUC0-last] | Up to 96hours
  The area under the concentration-time curve from time zero (pre-dose) to last time.
Pharmacokinetic parameters of SHR2150, , main metabolite and identified major metabolites in plasma ： [AUC0-∞] | Up to 96hours
  The area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time.
Pharmacokinetic parameters of SHR2150, , main metabolite and identified major metabolites in plasma ：[t1/2] | Up to 96hours
  Terminal Half-life
Pharmacokinetic parameters of SHR2150, , main metabolite and identified major metabolites in plasma： [Tmax] | Up to 96hours
  Time to Maximum Observed Concentration
Pharmacokinetic parameters of SHR2150, , main metabolite and identified major metabolites in plasma ： [Cmax] | Up to 96hours
  Maximum Observed Plasma Concentration
Pharmacokinetic parameters of SHR2150, , main metabolite and identified major metabolites in plasma ： [CL/F] | Up to 96hours
  Apparent clearance
Pharmacokinetic parameters of SHR2150, , main metabolite and identified major metabolites in plasma ： [Vz/F] | Up to 96hours
  Apparent volume of distribution
Pharmacokinetic parameters of SHR2150, , main metabolite and identified major metabolites in plasma ： [MRT] | Up to 96hours
  Mean retention time
Pharmacodynamics: Changes in Cytokines in Serum: interferon γ-inducible protein-10 | Up to 48hhours
Pharmacodynamics: Changes in Cytokines in Serum: Interferon-α | Up to 48hours

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing youan Hospital,Capital medical university, Beijing, Beijing Municipality, China